CLINICAL TRIAL: NCT00066248
Title: The Effect of Cyproheptadine Hydrochloride (Periactin) and Megestrol Acetate (Megace) on Weight in Children With Cancer/Treatment Related Cachexia
Brief Title: Cyproheptadine and Megestrol in Preventing Weight Loss in Children With Cachexia Caused By Cancer or Cancer Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: SCUSF 0205; HLMCC-0205 (Other: H. Lee Moffitt Cancer Center Research Base); U10CA081920 (NIH); SCUSF 0205 (Other: SunCoast CCOP Research Base)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Brain Tumor; Central Nervous System Tumors; Cachexia; Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: cachexia; unspecified childhood solid tumor; childhood spinal cord neoplasm; recurrent childhood medulloblastoma; untreated childhood medulloblastoma; childhood high-grade cerebral astrocytoma; childhood low-grade cerebral astrocytoma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; untreated childhood cerebellar astrocytoma; childhood oligodendroglioma; recurrent childhood brain stem glioma; recurrent childhood visual pathway glioma; hypothalamic glioma; untreated childhood brain stem glioma; untreated childhood visual pathway; childhood supratentorial primitive neuroectodermal tumor; childhood craniopharyngioma; childhood infratentorial ependymoma; childhood supratentorial ependymoma; newly diagnosed childhood ependymoma; recurrent childhood ependymoma; childhood choroid plexus tumor; childhood central nervous system germ cell tumor; childhood acute lymphoblastic leukemia in remission; recurrent childhood acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia; childhood acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia; untreated childhood acute myeloid leukemia; other myeloid malignancies; refractory chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; juvenile myelomonocytic leukemia; recurrent/refractory childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage II childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; untreated hairy cell leukemia; recurrent childhood lymphoblastic lymphoma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; stage I childhood small noncleaved cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; stage I childhood large cell lymphoma; stage II childhood large cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood brain tumor; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease; childhood chronic myelogenous leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; chronic myelomonocytic leukemia
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms; Cachexia; Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Spinal Cord Neoplasms; Medulloblastoma; Astrocytoma; Oligodendroglioma; Optic Nerve Glioma; Familial ependymoma; Choroid Plexus Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Recurrence; Leukemia, Hairy Cell; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Chronic | interventions — Cyproheptadine; Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subjects that respond to Periactin (Experimental): Receive 0.25mg/kg cyproheptadine hydrochloride once daily for 4 weeks. If subject responds to treatment (stable or increased weigh), go off study. If subject does not respond (loses weigh), subject will switch to10 mg/lg/day of megestrol acetate for 4 weeks.
  Interventions: Drug: cyproheptadine hydrochloride
- Non-responders to Periactin- Megace Arm (Experimental): Receive 0.25mg/kg cyproheptadine hydrochloride once daily for 4 weeks. If subject responds to treatment (stable or increased weigh), go off study. If subject does not respond (loses weigh), subject will switch to10 mg/lg/day of megestrol acetate for 4 weeks.
  Interventions: Drug: cyproheptadine hydrochloride; Drug: megestrol acetate

INTERVENTIONS:
Drug: cyproheptadine hydrochloride — Receive 0.25mg/kg cyproheptadine hydrochloride once daily for 4 weeks. If subject responds to treatment (stable or increased weigh), go off study. If subject does not respond (loses weigh), subject will switch to10 mg/lg/day of megestrol acetate for 4 weeks.
  Other Names: Periactin
Drug: megestrol acetate — Receive 0.25mg/kg cyproheptadine hydrochloride once daily for 4 weeks. If subject responds to treatment (stable or increased weigh), go off study. If subject does not respond (loses weigh), subject will switch to10 mg/lg/day of megestrol acetate for 4 weeks.
  Other Names: Megace
  Arms: Non-responders to Periactin- Megace Arm

SUMMARY:
RATIONALE: Cyproheptadine and megestrol may improve appetite and help prevent weight loss in children with cancer.

PURPOSE: This phase II trial is studying how well cyproheptadine and megestrol work in improving appetite and preventing weight loss in children with cachexia caused by cancer or cancer treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of cyproheptadine in preventing further weight loss in children with cancer or cancer treatment-related cachexia.
* Determine the efficacy of megestrol in preventing further weight loss in patients who don't respond to cyproheptadine.
* Determine how these drugs affect body protein and fat levels in these patients.

OUTLINE: Patients receive oral cyproheptadine twice daily for 4 weeks in the absence of unacceptable weight loss or toxicity. Patients that present with weight loss after 4 weeks receive oral megestrol daily for 4 weeks in the absence of unacceptable weight loss or toxicity. Patients responding to either cyproheptadine or megestrol may continue treatment at the discretion of the treating physician.

Patients are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 70 patients will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Any cachectic patient with weight loss presumed secondary to cancer or cancer related therapy is eligible. Cachexia is defined as having one or more of the following:
* documented history of weight loss > 5%
* drop in growth rate two or more percentile ranks on standard growth charts,
* weight for height less than the tenth percentile.
* Patients with newly diagnosed or relapsed cancer of any type, including brain tumors.
* Patients who are receiving active or palliative therapy are eligible.
* If patients have completed treatment for cancer (surgery, chemotherapy, radiotherapy) within 8 weeks of study registration, they are also eligible.
* Patients must be ≥ 2 years and < 21 years of age at the time of admission to this study.
* Patients must have a predicted life expectancy of at least eight weeks.

EXCLUSION CRITERIA:

* Patients who are currently taking or who have taken Periactin and/or Megace during the past three weeks are not eligible.
* Patients receiving corticosteroid or monoamine oxidase (MAO) inhibitor therapy. (Intermittent steroid use is permitted IF you anticipate it will not be administered for more than 7 days in a 4 week period. Calculate anticipated intermittent steroid use in 4-week intervals through the 8-week period during which study agent may be administered (4 weeks for Periactin and potentially 4 weeks for Megace.
* Patients who have received parenteral nutrition or tube feedings within 1 week of starting this protocol or patients who are expected to require parenteral nutrition or tube feedings during the 4-week course of this study.
* Patients taking dronabinol (Marinol) or other appetite-stimulating medications during the past three weeks or patients expected to be prescribed appetite-stimulating medications during the 4-week course of this study.
* Patients with hormone sensitive tumors specifically meningiomas, breast cancer, ovarian cancer, and endometrial carcinoma.31, 32
* Children with neurofibromatosis, type I or II, are at risk for the development of meningiomas and are thus excluded from this study.32
* Children with glaucoma, chronic persistent asthma, or gastrointestinal (GI) or genitourinary (GU) obstruction.
* Patients with recurrent and/or persistent hypertension, defined as blood pressure values >20% above normal.
* Patients with thromboembolic disease, congestive heart failure, or peripheral edema.
* Patients who are pregnant.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2003-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Efficacy of study agents as measured by changes in weight at baseline, and 4 weeks after the beginning of study treatment | 4-8 weeks

SECONDARY OUTCOMES:
Effect of study agents on protein and fat levels as measured by pre-albumin and lipid profile at baseline, and 4 weeks after the beginning of study treatment | 4-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L. Mayer, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (43):
- United States (40):
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Children's Hospital & Research Center Oakland, Oakland, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Children's Hospital of Tampa, Tampa, Florida
  - CCOP - Florida Pediatric, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Floating Hospital for Children at Tufts - New England Medical Center, Boston, Massachusetts
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Detroit, Michigan
  - DeVos Children's Hospital, Grand Rapids, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Saint Paul, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Tomorrows Children's Institute at Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Tod Children's Hospital, Youngstown, Ohio
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - CHRISTUS Santa Rosa Children's Hospital, San Antonio, Texas
  - MBCCOP - South Texas Pediatrics, San Antonio, Texas
  - Methodist Cancer Center at Methodist Specialty and Transplant Hospital, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
- Canada (2):
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
- San Jorge Children's Hospital, Santurce, Puerto Rico

REFERENCES:
- [Result] Couluris M, Mayer JL, Freyer DR, Sandler E, Xu P, Krischer JP. The effect of cyproheptadine hydrochloride (periactin) and megestrol acetate (megace) on weight in children with cancer/treatment-related cachexia. J Pediatr Hematol Oncol. 2008 Nov;30(11):791-7. doi: 10.1097/MPH.0b013e3181864a5e. PMID 18989154